CLINICAL TRIAL: NCT04077554
Title: Relationship Between the VEGF Gene Polymorphism and Cardiometabolic Risk Factors in People With Excessive Body Weight in the Polish Population
Brief Title: Relationship Between the VEGF Gene Polymorphism and Cardiometabolic Risk Factors
Acronym: 27/MN/2018
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Damian Skrypnik, MD, PhD, Principial Investigator, Poznan University of Medical Sciences
Other Study IDs: 359/15 & 1309/18
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Polymorphism, Restriction Fragment Length
Keywords: VEGF gene expression; VEGF gene polymorphism; leptin
MeSH Terms: interventions — Gene Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — salting out method was developed from blood and DNA was protected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: women and men with excess body mass
  Interventions: Genetic: gene expression
- Control group: women and men with proper body mass
  Interventions: Genetic: gene expression

INTERVENTIONS:
Genetic: gene expression — determination of VEGF gene expression, VEGF gene polymorphism and serum leptin concentration

SUMMARY:
The aim of the study is to determine the relationship between VEGF gene expression, VEGF gene polymorphism and serum leptin concentration in the Polish population in people with excessive body weight. In addition, the aim of the study is to look for relationships between the VEGF gene polymorphism and anthropometric and biochemical factors of cardiovascular risk and endothelial dysfunction such as body weight, waist circumference, serum total cholesterol, LDL, HDL, triglycerides, glucose and the occurrence of cardiovascular diseases in the family of a patient with excessive body weight in the Polish population.

DETAILED DESCRIPTION:
400 people (250 - study group; 150 control group) were subjected to subjective and objective action. Information on the occurrence of diseases and cardiovascular risk in the participant and his family was collected from research studies. Anthropometric parameters were measured (body weight, height, BMI, waist circumference, neck circumference) as well as blood pressure and pulse measurement. In addition, fasting venous blood was collected and secured. In venous blood currently marked with the following concentration: glucose, required cholesterol, LDL cholesterol, HDL cholesterol and triglycerides. In addition, a method of salting out and protecting DNA was developed from blood.

Furthermore the polymorphisms of VEGF genes (in positions: -2578 and -634) using the HMR (High Resolution Melt) method was determined.

Also VEGF and leptin by ELISA was determined. After obtaining the results of comparative analysis of the correlation between the occurrence of VEGF gene polymorphisms, serum levels of leptin and VEGF, and anthropometric and biochemical parameters of cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* informed consent in writing
* stable body mass (+/- 1 kg)
* excessive body mass (BMI ≥ 25 kg/m2- study group)
* proper body mass (BMI < 25 kg/m2- control group)

Exclusion Criteria:

* age <18 years
* secondary obesity
* pregnancy, lactation
* other conditions that in the opinion of researchers may pose any risk to the patient during the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 195/5000 250 people (women and men) with excessive body weight (BMI ≥ 25 kg / m2 - study group) and 150 people (women and men) with normal body weight (BMI <25 kg / m2 - control group) from Poland.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
VEGF gene expression | through study completion, an average of 1 year
  VEGF gene expression
VEGF gene polymorphism | through study completion, an average of 1 year
  VEGF gene polymorphism
serum leptin concentration | through study completion, an average of 1 year
  serum leptin concentration

SECONDARY OUTCOMES:
Body mass (BM) | through study completion, an average of 1 year
  Body mass
Waist circumference (WC) | through study completion, an average of 1 year
  Waist circumference
total cholesterol (TCH) | through study completion, an average of 1 year
  Blood concentration of total cholesterol
low density lipoprotein (LDL) | through study completion, an average of 1 year
  Blood concentration of low density lipoprotein
high density lipoprotein (HDL) | through study completion, an average of 1 year
  Blood concentration of high density lipoprotein
triglycerides | through study completion, an average of 1 year
  Blood concentration of triglycerides
glucose | through study completion, an average of 1 year
  Blood concentration of glucose

CONTACTS AND LOCATIONS:
Overall Officials: Damian Skrypnik, MD; PhD, Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Department of Treatment of Obesity, Metabolic Disorders and Clinical Dietetics, Poznan University of Medical Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skrypnik D, Mostowska A, Jagodzinski PP, Bogdanski P. Association of rs699947 (-2578 C/A) and rs2010963 (-634 G/C) Single Nucleotide Polymorphisms of the VEGF Gene, VEGF-A and Leptin Serum Level, and Cardiovascular Risk in Patients with Excess Body Mass: A Case-Control Study. J Clin Med. 2020 Feb 8;9(2):469. doi: 10.3390/jcm9020469. PMID 32046348